CLINICAL TRIAL: NCT01184443
Title: Evaluation of the Efficacy and Safety of Olanzapine as an Adjunctive Treatment for Anorexia Nervosa in Children and Adolescents: An Open-label Trial
Brief Title: Evaluation of the Efficacy and Safety of Olanzapine for Anorexia Nervosa in Children and Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Wendy Spettigue, MD, FRCPC, Child and Adolescent Psychiatrist, Children's Hospital of Eastern Ontario
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGDM24
Record Dates: First submitted 2010-08-13; First posted 2010-08-19 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Eating Disorder
Keywords: Anorexia Nervosa; Eating Disorder Not Otherwise Specified; Olanzapine; Pediatric
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine (Experimental): Those who choose to take olanzapine as part of their treatment (standard practice plus medication).
  Interventions: Drug: Olanzapine
- Comparison (No Intervention): Those who choose not to take olanzapine as part of their treatment (standard practice).

INTERVENTIONS:
Drug: Olanzapine — Dosing regimen is in keeping with clinical practice. Patients will typically start oral olanzapine at 2.5mg (rarely 1.25mg) daily for 1 to 2 weeks, and if tolerated and clinically indicated, are increased to 5.0mg daily. The majority of patients will remain on a maintenance dose of 5.0mg, but more agitated patients may take 7.5mg (rarely 10.0mg) daily. Patients will be tapered off as they approach/attain their ideal body weight.
  Other Names: Teva-Olanzapine; Dins: 02276712 and 02276720
  Arms: Olanzapine

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of the atypical antipsychotic, olanzapine, for the treatment of youth suffering from Anorexia Nervosa (AN).

Adolescent males and females between the ages of 11 and 17 years who are being treated by a physician on the Eating Disorder team at the Children's Hospital of Eastern Ontario will be invited to join the study if they have been diagnosed with AN or Eating Disorder Not Otherwise Specified (EDNOS), and if they weigh less than or equal to 85% of their ideal body weight. Those who meet inclusion and not exclusion criteria, and consent to participating in the trial will be offered adjunctive treatment with olanzapine. Those who agree to take olanzapine will belong to the olanzapine group, and those who decline will belong to the comparison group. Olanzapine doses will be in keeping with the investigators current clinical practice, with flex doses ranging from 1.25 mg to 10.0 mg daily (the majority of patients are treated with 2.5 mg or 5.0 mg at bedtime); dose adjustments made based on individual need and tolerability. Participants will remain in the study for 12 weeks. Those who initially decline olanzapine treatment may change their minds and take olanzapine up until week 9 of the trial.

It is hypothesized that those children and adolescents who choose to take olanzapine at entry into the trial will be more motivated to recover and more compliant with treatment. Compared to those who do not receive medication, it is expected that these adolescents will demonstrate reduced disordered eating attitudes and behaviours, as well as an increased rate of weight gain.

Finally, it is predicted that the rates of discontinuation and the adverse effects of olanzapine will be minor given the relatively low dose (as compared to treatment for patients with schizophrenia), slow titration, and short-term use of olanzapine the investigators will be using.

By comparing the well-being and outcome of patients in the two groups, the investigators hope to begin to answer the question of whether olanzapine does or does not lead to improved clinical outcome for patients with severe eating disorders such as AN or EDNOS, and the question of whether the benefits of using the medication outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 11 and 17 (less than 18) at beginning of trial
* Based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), patient fulfills criteria for diagnosis of Anorexia Nervosa (of which there are two types: restricting or binge-eating/purging) or Eating Disorder Not Otherwise Specified, with a weight of less than or equal to 85% of his or her ideal body weight, as can best be determined at the time of assessment
* Treated by physician on the eating disorder team at the Children's Hospital of Eastern Ontario (CHEO)

Exclusion Criteria:

* Currently receiving treatment with any other antipsychotic medication, mood stabiliser, or stimulant
* Known diagnosis of: diabetes, impaired glucose tolerance, hyperlipidemia, hepatic dysfunction, substance dependence, narrow angle glaucoma, paralytic ileus, or pancreatitis, or any other medical illness that would be considered to significantly impact treatment or recovery from the eating disorder
* Any uncontrolled comorbid disease affecting any system including infectious, endocrine, renal, gastroenterologic, respiratory, cardiac, immunologic, or hematologic. Potential participants with controlled comorbidities in these areas may be invited to participate at the discretion of the primary investigator.
* Experienced one or more seizures without clear and resolved etiology
* Inability to comply with trial requirements including lack of comprehension of English
* Pregnant or breast-feeding
* High blood pressure
* Known allergy or known sensitivity to products in olanzapine
* Other unspecified reasons that, in the opinion of the investigator, amke the patient unsuitable for enrollment
* Officially declared incapable of consenting to treatment under the Mental Health Act (Note: If a patient is involuntarily hospitalized, he or she can be invited to participate provided that he or she has not officially been deemed incapable of making treatment decision under the Mental Health Act)
* Clinically judged to be at serious suicidal ris
* More than 6 months have passed between the patient's initial eating disorder assessment and the time of study entry
* Liver function test (ALT) > 1.5 x upper limit of normal (ULN)
* Positive pregnancy test
* Electrocardiogram (ECG): QTc > 450 msec or arrythmia other than sinus bradycardia; conduction abnormalities, prolonged QTc or other
* LDL-C > 4.9 mmol/L
* Total cholesterol/HDL ratio > 6
* Fasting glucose > or equal to 6.1 mmol/L
* Neutrophil count < 0.5 x 10^9/L
* Prolactin level at assessment > 200 ng/mL

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Symptom Severity Scale | 12 weeks
  Psychological Primary Outcome: The Eating Disorder Symptom Severity Scale is a clinician-rated measure of eating disorder severity, and behavioural and cognitive eating disorder symptoms.
Rate of weight gain | 12 weeks
  Medical Primary Outcome: Rate of weight gain will be measured throughout the trial.

SECONDARY OUTCOMES:
Children's Depression Inventory | 12 weeks
  Psychological measure that assesses cognitive, behavioural, and somatic symptoms of depression.
Multidimensional Anxiety Scale for Children | 12 weeks
  Psychological measure that assesses anxiety.
Eating Disorder Examination Questionnaire-Adolescent | 12 weeks
  Assesses behaviours and attitudes associated with eating disorders in youth 13 years of age and older.
The Children's Eating Attitudes Test | 12 weeks
  Assesses behaviours and attitudes associated with eating disorders in youth between the ages of 8 and 12.
Child Behavior Checklist | 12 weeks
  Evaluates parents' perceptions of their child's mood and anxiety
Eating Disorder Restlessness Agitation Drug Sleep Scale (for youth and parents) | 12 weeks
  Thes questionnaire asks specific questions about restlessness, eating disorder cognitions, sleep, medication, and the patient's desire to recover from the eating disorder, that are not addressed in the other questionnaires.
Eating Disorder Inventory-3 | 12 weeks
  Psychological measure that assess psychological traits and symptoms relevant to the development and maintenance of eating disorders.
Overall Safety Profile | 12 weeks
  An overall assessment of the safety profile of olanzapine will be done. This will include examination of reported adverse events, vital signs, electrocardiograms, urinalysis, and blood chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Spettigue, MD, FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Spettigue W, Norris ML, Maras D, Obeid N, Feder S, Harrison ME, Gomez R, Fu MC, Henderson K, Buchholz A. Evaluation of the Effectiveness and Safety of Olanzapine as an Adjunctive Treatment for Anorexia Nervosa in Adolescents: An Open-Label Trial. J Can Acad Child Adolesc Psychiatry. 2018 Aug;27(3):197-208. Epub 2018 Jul 1. PMID 30038658